CLINICAL TRIAL: NCT02079311
Title: Evaluation of Perioperative Core Body Temperature When Using Forced Air Warming or BARRIER® EasyWarm to Prevent Inadvertent Perioperative Hypothermia: An Open-label, Randomized Non-inferiority Comparison
Brief Title: Evaluation of Core Body Temperature When Using Forced Air Warming or an Active Blanket to Prevent Perioperative Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD13-001
Record Dates: First submitted 2014-02-18; First posted 2014-03-05 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2014-06

CONDITIONS: Inadvertent Perioperative Hypothermia; Preoperative Anxiety Experienced by the Patient
Keywords: Patient warming; Active warming; Forced Air Warming; Warming blanket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active self-warming blanket (Experimental): Active warming with BARRIER® EasyWarm active self-warming blanket during the perioperative phase
  Interventions: Device: Active self warming blanket
- Forced air warming device (Active Comparator): Active warming with forced air warming (FAW) during the intraoperative phase.
  Interventions: Device: Forced air warming device

INTERVENTIONS:
Device: Active self warming blanket — BARRIER® EasyWarm is a disposable self-warming blanket that produces heat via an exothermic chemical reaction initiated by exposure to air, resulting from the oxidation of iron.
  Other Names: BARRIER® EasyWarm
  Arms: Active self-warming blanket
Device: Forced air warming device — Forced air warming is a temperature management unit, where heated air is used to warm subjects through convection.
  Other Names: Bair Hugger™; Equator® level 1.
  Arms: Forced air warming device

SUMMARY:
This investigation is undertaken to investigate if patient warming with BARRIER® EasyWarm active self-warming blanket differs compared to active warming with forced air warming in terms of core body temperature perioperatively.

A non-inferiority, prospective, open-labelled, randomized, parallel investigation.

Randomized subjects will receive active warming with BARRIER® EasyWarm or with forced air warming. All subjects may receive rescue warming if their core temperature falls below 35.5°C. Rescue warming is optional and defined as the institution's standard of care to prevent hypothermia.

The primary purpose is to investigate if there is a clinically relevant difference in core body temperature between the two treatment groups.

A total of 60 subjects will be included in the investigation, i.e. 30 subjects in each treatment group. The number includes a 30% drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent i.e. subject must be able to understand and sign the Informed Consent Form (ICF)
* Male and female subjects aged 18 years and over
* Subject scheduled for surgery with a minimum length of 60 minutes and a maximum length of 120 minutes
* Scheduled surgery must be performed entirely under general anaesthesia
* The subject must be able to receive temperature assessments via an oesophageal temperature probe when under general anaesthesia and via an oral thermometer before and after general anaesthesia as well as in the pre- and post-op area
* The subject must have an oral temperature measurement of at least 36.0°C when first measured in the preoperative setting
* The subject's scheduled surgical procedure must allow time to be warmed with a fully activated BARRIER® EasyWarm at least 30 minutes prior to induction of general anaesthesia

Exclusion Criteria:

* Subjects with an American Society of Anesthesiologists (ASA) rating of 4 or greater
* Known Diabetes with an HbA1c of more than 6 %
* Relevant medical history (e.g., neuropathy, peripheral vascular disease, circulatory disorder or other) that presents risk to/of:

  1. The subject's normal temperature regulation or
  2. Perception of external temperature or
  3. Subcutaneous lipoatrophy
* Current use of concomitant medications that present relevant risk to/of:

  1. The subject's normal temperature regulation or
  2. Perception of external temperature or
  3. Subcutaneous lipoatrophy
* Epidural/Spinal anaesthesia
* An oral temperature measurement ≥ 37.5°
* Contraindications to the oesophagus temperature probe and oral thermometer
* Presence of skin and soft tissue disorders in areas covered directly by the device in the two treatment groups (e.g. pressure ulcers, clinically significant psoriasis, dermatitis or any other interruption of skin integrity that would be affected by direct heat)
* Pregnancy
* Severe non-compliance to protocol as judged by the investigator and/or Mölnlycke Health Care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Torossian, Prof. MD, Principal Investigator — Universitätsklinikum Gießen und Marburg GmbH
Locations (3):
- Universitätsklinikum Gießen und Marburg GmbH, Marburg, Germany
- Ullevål - Oslo Universitetssykehus, Oslo, Norway
- Royal Hallamshire Hospital, Sheffield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Self-warming Blanket | Forced Air Warming Device
Started | 28 | 27
Completed | 28 | 26
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Self-warming Blanket | Forced Air Warming Device | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 49 (13.2) | 50 (14.44) | 49.5 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants] — 2 subject were enrolled but not randomised.
  participants
    Germany | 15 | 14 | 29
    Norway | 7 | 7 | 14
    United Kingdom | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Core Body Temperature in the Two Treatment Groups.
Description: Temperature assessments will be made using an oesophageal temperature probe when the subject is under general anaesthesia and by oral thermometer for all other temperature assessments performed in pre-, intra- and post-op. The mean value is calculated on all temperature measured during pre-, intra- and post-op.
Time Frame: Subjects will be followed for one day of hospital stay, data to be collected during the perioperative phase. Expected to be between 5-8 hours.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Active Self-warming Blanket | Forced Air Warming Device
Number analyzed (Participants) | 28 | 27
degree celsius | 36.28 (0.3) | 36.25 (0.33)

ADVERSE EVENTS:
Arm/Group | Active Self-warming Blanket | Forced Air Warming Device
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 12/28 | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Self-warming Blanket (N=28) | Forced Air Warming Device (N=27)
redness (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1) — redness of skin vanished quickly without treatment
hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Hematoma on the left gluteus maximus and the right knee. Not related to investigational product.
anaphylactic shock (Vascular disorders) | 0 (0) | 1 (1) — Anaphylactic shock due to blue methylene intracutan injection. The subject was planned to have a breast surgery due to cancer mammae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall provide the Sponsor with a draft of the manuscript intended for publication or presentation at least [14] days before the date of intended submission for publication. However the Sponsor should be notified about the intention to publish the results at least [14] days before the manuscript is sent for review. All comments and suggested changes made by the Sponsor shall be considered in good faith in determining the final form of such publication.